CLINICAL TRIAL: NCT06565975
Title: RELION Study: Characteristics and Outcomes of the Patient Population With Acute Myeloid Leukemia in Remission, Treated With Oral Azacitidine Maintenance in France
Brief Title: Characteristics and Outcomes of Acute Myeloid Leukemia (AML) Patients Treated With Oral-Azacitidine Maintenance Therapy in France
Acronym: RELION
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA055-1047
Record Dates: First submitted 2024-07-22; First posted 2024-08-22 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: Acute myeloid leukemia (AML)
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants that received maintenance treatment of oral azacitidine
  Interventions: Drug: Oral azacitidine

INTERVENTIONS:
Drug: Oral azacitidine — As per product label, prescribed by treating physician

SUMMARY:
The purpose of this study is to collect and evaluate real-world data to describe the outcomes, patient characteristics, safety profile and treatment patterns of oral azacitidine prescribed as maintenance treatment after frontline treatment or second remission for acute myeloid leukemia in France.

ELIGIBILITY:
Inclusion Criteria:

* Participants who initiated oral azacitidine maintenance therapy during early access program (EAP) in France (January 29, 2021 to July 13, 2022) or during the 6 months post-EAP (from July 14, 2022, to January 2014, 2023) inside the marketing authorization label "adult patients with acute myeloid leukaemia (AML) who achieved complete remission (CR) or complete remission with incomplete blood count recovery (CRi) following induction therapy with or without consolidation treatment and who are not candidates for, including those who choose not to proceed to, hematopoietic stem cell transplantation (HSCT)."
* Participants with histologically confirmed diagnosis of de novo AML, or therapy-related AML, or secondary AML
* Participants who received frontline treatment after diagnosis of AML and achieved complete remission (CR), CR with incomplete blood count recovery (Cri), or CR with partial hematology recovery (CRh) after one or subsequent lines of therapy in case of relapse
* Participant is at least 18 years of age at the time of initial diagnosis of AML
* Participants alive or deceased at the time of data collection
* Physician has access to the complete medical record for the patient, including any transferred records from other facilities (if applicable); patient's medical record must at least include the following:

  * Date of diagnosis of AML
  * Frontline therapy(ies) received, and treatment start dates
  * Date(s) of first documented evidence of response
  * Oral azacitidine start and (if applicable) stop date
  * Documentation (yes/no) of relapse on oral azacitidine, where applicable
* Participants who do not object to the data collection

Exclusion Criteria:

* Participants who initiated maintenance with oral azacitidine after January 14, 2023
* Participant who initiated maintenance with oral azacitidine before January 14, 2023, outside of the marketing authorization label

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with histologically confirmed de novo acute myeloid leukemia, therapy-related acute myeloid leukemia, or secondary acute myeloid leukemia who received maintenance therapy with oral azacitidine while in remission after front-line treatment or in second remission
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2026-01-26 (Actual); Study Completion 2026-01-26 (Actual)

PRIMARY OUTCOMES:
Participant real-world relapse-free survival (rw-RFS) | Up to date of documented relapse or death assessed up to 41 months
Participant overall survival (OS) | Up to date of documented death assessed up to 41 months
Participant relapsed-free survival (RFS) | From date of achieved complete remission up to 41 months
Participant overall survival (OS) from the time of complete remission achievement | From date of achieved complete remission up to 41 months
Participant relapse rate | 6 and 12 months
Time to treatment discontinuation (TTD) | Up to 41 months

SECONDARY OUTCOMES:
Participant baseline demographics | Baseline
Type of acute myeloid (AML) | Baseline
  AML types include: de novo, or secondary AML (therapy-related AML, or secondary to a myeloid disorder)
Participant cytogenetic abnomalities | Baseline
Participant gene mutation status | Baseline
Participant cytogenetic and mutational risk category | Baseline
Participant acute myeloid (AML) classification as per World Health Organization | Baseline
Participant bone marrow blast percentage | Baseline
Participant hemoglobin levels | Baseline
Participant blood test results | Baseline
Participant Eastern Cooperative Oncology Group or Karnofsky score | Baseline
Participant diagnosis history of other hematological disorders | Baseline
Participant treatment history | Baseline
Minimal residual disease status (MRD) | Baseline
Reason for stem cell transplant ineligibility post initial frontline treatment | Baseline
Participant response type at the initiation of maintenance therapy | Up to 41 months
  Response types include: complete remission (CR), incomplete blood count recovery (Cri) or CR with partial hematology recovery (CRh)
First versus subsequent remission at the time of initiation of treatment with oral azacitidine | Baseline
Criteria to define complete remission (CR), incomplete blood count recovery (Cri), and CR with partial hematology recovery (CRh) at time of initiation of oral azacitidine | Baseline
Oral azacitidine treatment regimen | Up to 41 months
Concomitant support treatment received with oral azacitidine | Up to 41 months
Duration of oral azacitidine treatment | Up to 41 months
Reason for oral azacitidine treatment discontinuation | Up to 41 months
Treatments/procedures following oral azacitidine cessation | Up to 41 months
Participant adverse events (AEs) | Up to 41 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Kappa Sante, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts